CLINICAL TRIAL: NCT06129123
Title: Development of An Online, Theory-Based Intervention to Reduce E-cigarette Use and Susceptibility to Smoking in Young Adults: A Pilot Study
Brief Title: An Online Intervention to Reduce E-cigarette Use and Susceptibility to Smoking in Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Denise Tran, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UP-23-00005-AM001
Record Dates: First submitted 2023-11-08; First posted 2023-11-13 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: E-cigarette Use
MeSH Terms: conditions — Vaping

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be asked to complete a 30-minute intervention that is accessible on a mobile device, delivered via a webpage, and personalized to their individual vaping behavior and beliefs (based on the baseline surveys). The intervention will contain personalized normative feedback (PNF), Motivational Enhancement (ME), and education.
  Participants will complete assessments at baseline as well as 2-weeks, 4-weeks, and 8-weeks post randomization.
  Interventions: Behavioral: Live Free From E-cigarettes
- Waitlist Control (No Intervention): Participants will complete assessments at baseline as well as 2-weeks, 4-weeks, and 8-weeks post randomization. They will not receive the intervention during the active study phase, lasting 8 weeks. Participants will have the option to access the intervention once this active study phase is over.

INTERVENTIONS:
Behavioral: Live Free From E-cigarettes — This is a 30-minute online educational program that focuses on providing information about e-cigarette and smoking social norms, harms of e-cigarettes and cigarettes, and ways to quit or reduce using e-cigarettes.
  Arms: Intervention

SUMMARY:
The goal of this intervention development and pilot clinical trial is to determine whether receiving the brief online intervention results in greater reductions in past 7-day e-cigarette use frequency and smoking susceptibility over an 8-week period compared to receiving the control condition in young adults who currently use e-cigarettes. Participants in the experimental condition will be asked to complete the 30-minute mobile-based program. Participants in the assessment-only control will be given the option to access the intervention after they complete their final survey at 8 weeks. All participants will complete our online surveys at baseline as well as 2-weeks, 4-weeks, and 8-weeks post-randomization. Researchers will compare outcomes among the intervention and control groups to determine the efficacy of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18 to 24
* be able to read English
* report vaping at least one day per week in the past month
* report no history of cigarette use at screening and baseline.

Exclusion Criteria:

* reporting severe mental health, illicit drug use, or alcohol use disorder
* currently receiving nicotine cessation services

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-01-23 (Estimated); Study Completion 2026-01-23 (Estimated)

PRIMARY OUTCOMES:
E-cigarette Use | 8 weeks
  Participants will report the number of (1) days they vaped, (2) times they picked up their device to vape per day, and (3) puffs they took before putting their vaping device away per day in the past 7 days and 30 days
Smoking Susceptibility | 8 weeks
  4-item Expanded Susceptibility to Smoking Index (ESSI)

SECONDARY OUTCOMES:
Perceived harms and benefits of vaping | 8 weeks
  Using the 21-item Short Form Vaping Consequences Questionnaire (S-VSQ), participants will rate the likelihood that each consequence will occur when they vape.
Perceived harms and benefits of smoking | 8 weeks
  Using the 21-item Short Form Smoking Consequences Questionnaire (S-SCQ), participants will rate the likelihood that each consequence will occur when they smoke.
Motivation to vape | 8 weeks
  Participants will select which option best describes their interest in e-cigarette use: plan to stop (coded as 1), decrease (2), continue (3) or increase (4) vaping.
Motivation to smoke | 8 weeks
  Participants will report if they plan to start smoking (yes/no).
Quitting vaping self-efficacy | 8 weeks
  Participants rate their confidence about quitting vaping "someday" and "in the next 6 months" on a 5-point scale.
Vaping quit attempts | 8 weeks
  During follow-up assessments, participants will report on the number of times they have stopped vaping for one day or longer because they were trying to quit vaping.

CONTACTS AND LOCATIONS:
Overall Officials: Denise D Tran, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No
No identifying participant information will be shared with other researchers. In the case where another researcher requests access to our data, we will de-identify our data set before sharing these data.

REFERENCES:
- [Derived] Tran DD, Davis JP, Buch K, Leventhal AM, Ewing SWF, Pedersen ER. A novel online vaping intervention and smoking prevention program for young adults who vape: protocol for a randomized controlled trial. Addict Sci Clin Pract. 2025 Apr 21;20(1):36. doi: 10.1186/s13722-025-00566-x. PMID 40259422